CLINICAL TRIAL: NCT05810727
Title: Temporal Changes in Clinical Characteristics and Functions, and Their Relationship With Outcomes of Atrial Fibrillation: a Retrospective Study Utilizing Data Linkage of a Single Center Patient Data and National Claims Database in Korea
Brief Title: Atrial Fibrillation Data Linkage Non-Interventional Study
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661188; Eliquis AF data linkage NIS (Other: Alias Study Number)
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to understand temporal changes in clinical features and functions, and the relationship with outcomes of atrial fibrillation (AF). AF is a problem with speed or pattern that the heart beats. It is the most common type of arrythmia. The study will use data linkage of a single center patient data and national claims database in Korea. This study does not include an actual patient enrollment process.

ELIGIBILITY:
Inclusion Criteria:

* Patients had incident AF diagnosis (International Classification of Diseases 10th Revision [ICD-10]; I48) in an inpatient or outpatient setting at SNUH between 1 Jan 2010 and 31 Dec 2020
* Patients aged 18 years or older on the index date

Exclusion Criteria:

* Medical claims indicating a diagnosis code indicative of rheumatic mitral valvular heart disease, mitral valve stenosis, or prosthetic heart valve during 12 months period prior to first AF diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients with Atrial Fibrillation diagnosis code at Seould National Universit Hospital(SNUH) from Jan 2010 to Dec 2020.
Sampling Method: Probability Sample
Enrollment: 12556 (Actual)
Dates: Start 2025-08-21 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Event Rate of Stroke/Systemic embolism (SE) | Up to 12 months after AF diagnosis or after the start date of relevant atrial fibrillation(AF) treatment
  National Health Insurance Service(NHIS)
  Claims with the following ICD-10 diagnosis codes as main or all sub-diagnoses whichever came first (i.e., the first occurred event will be used):
  1. Ischemic stroke: G45.9, I63, I69.3
  2. Hemorragic stroke: I60, I61, I62, I69.0, I69.1, I69.2
  3. Systemic embolism: I74
     * Hospitalization and computed tomography (CT) or magnetic resonance imaging (MRI) codes (brain CT or MRI for ischemic stroke and hemorrhagic stroke; any CT or MRI for systemic embolism) were also required for identification.
Event Rate of Major bleeding | Up to 12 months after the AF diagnosis or after the start date of relevant AF treatment
  Bleeding requiring hospitalization will be identified using hospital claims which had a bleeding diagnosis code as the first occurred ICD-10 code and will be consisted of intracranial hemorrahge (ICH), gastrointestinal (GI) bleeding, and other bleeding. Main and all sub-diagnosis codes will be used. Particularly, hospitalization and brain CT or MRI codes (as described in variable 'stroke or SE') will be needed to identify ICH.
All-Cause Mortality Rates | Up to 12 months after the AF diagnosis or after the start date of relevant AF treatment
  Death will be identified from mortality registration data of Statistics Korea linked to NHIS database

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661188